CLINICAL TRIAL: NCT05845671
Title: A Phase 1 / 2, Open Label, Study of Amivantamab (JNJ-61186372) Among Participants With Advanced NSCLC Harboring ALK, ROS1, and RET Gene Fusions in Combination With Tyrosine Kinase Inhibitors
Brief Title: Amivantamab With Tyrosine Kinase Inhibitors (TKI) for Advanced NSCLC With ALK, ROS1, or RET Alterations
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-1450.cc; 61186372LUC2005 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer
Keywords: ALK; ROS1; RET
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Finding (Safety Lead-In) Cohort (<80 kg) (Experimental): To estimate the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) in adult participants with advanced NSCLC with ALK, ROS1, and RET gene fusions.
  Interventions: Drug: Amivantamab 1050mg
- Dose Finding (Safety Lead-In) Cohort (≥80 kg) (Experimental): To estimate the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) in adult participants with advanced NSCLC with ALK, ROS1, and RET gene fusions.
  Interventions: Drug: Amivantamab 1400mg
- Dose Expansion Cohort (<80 kg) (Experimental): To estimate the objective response rate (ORR) of amivantamab in combination with common TKIs used in ALK, ROS1, and RET advanced NSCLC progressing on TKIs.
  Interventions: Drug: Amivantamab (to be determined)
- Dose Expansion Cohort (≥80 kg) (Experimental): To estimate the objective response rate (ORR) of amivantamab in combination with common TKIs used in ALK, ROS1, and RET advanced NSCLC progressing on TKIs.
  Interventions: Drug: Amivantamab (to be determined)

INTERVENTIONS:
Drug: Amivantamab 1050mg — Amivantamab is a bispecific antibody that binds to the extracellular domains of EGFR and MET.
  In in vitro and in vivo studies amivantamab was able to disrupt EGFR and MET signaling functions through blocking ligand binding and, in exon 20 insertion mutation models, degradation of EGFR and MET. The presence of EGFR and MET on the surface of tumor cells also allows for targeting of these cells for destruction by immune effector cells, such as natural killer cells and macrophages, through antibody-dependent cellular cytotoxicity (ADCC) and trogocytosis mechanisms, respectively.
  Other Names: JNJ-61186372
  Arms: Dose Finding (Safety Lead-In) Cohort (<80 kg)
Drug: Amivantamab 1400mg — Amivantamab is a bispecific antibody that binds to the extracellular domains of EGFR and MET.
  In in vitro and in vivo studies amivantamab was able to disrupt EGFR and MET signaling functions through blocking ligand binding and, in exon 20 insertion mutation models, degradation of EGFR and MET. The presence of EGFR and MET on the surface of tumor cells also allows for targeting of these cells for destruction by immune effector cells, such as natural killer cells and macrophages, through antibody-dependent cellular cytotoxicity (ADCC) and trogocytosis mechanisms, respectively.
  Other Names: JNJ-61186372
  Arms: Dose Finding (Safety Lead-In) Cohort (≥80 kg)
Drug: Amivantamab (to be determined) — Amivantamab is a bispecific antibody that binds to the extracellular domains of EGFR and MET.
  In in vitro and in vivo studies amivantamab was able to disrupt EGFR and MET signaling functions through blocking ligand binding and, in exon 20 insertion mutation models, degradation of EGFR and MET. The presence of EGFR and MET on the surface of tumor cells also allows for targeting of these cells for destruction by immune effector cells, such as natural killer cells and macrophages, through antibody-dependent cellular cytotoxicity (ADCC) and trogocytosis mechanisms, respectively.
  Dose will be determine after the Safety Lead-In
  Other Names: JNJ-61186372
  Arms: Dose Expansion Cohort (<80 kg)
Drug: Amivantamab (to be determined) — Amivantamab is a bispecific antibody that binds to the extracellular domains of EGFR and MET.
  In in vitro and in vivo studies amivantamab was able to disrupt EGFR and MET signaling functions through blocking ligand binding and, in exon 20 insertion mutation models, degradation of EGFR and MET. The presence of EGFR and MET on the surface of tumor cells also allows for targeting of these cells for destruction by immune effector cells, such as natural killer cells and macrophages, through antibody-dependent cellular cytotoxicity (ADCC) and trogocytosis mechanisms, respectively.
  Dose will be determine after the Safety Lead-In
  Other Names: JNJ-61186372
  Arms: Dose Expansion Cohort (≥80 kg)

SUMMARY:
Although non-small cell lung cancer (NSCLC) patients with anaplastic lymphoma kinase (ALK), c-ros oncogene 1(ROS1), and ret proto-oncogene (RET) gene fusions initially respond well to tyrosine kinase inhibitor (TKI) therapies, acquired resistance is inevitable. In many of these cases, increased activation of the erythroblastic leukemia viral oncogene homologue (ERBB) or cMet pathways appears to be a bypass signaling mechanism that allows these cancer cells to circumvent the selective pressure from TKIs. Recent data have suggested that these pathways compensate for each other in situations where one pathway is inhibited, leading to "kinase switch" drug resistance. Thus, the expected inhibition of both pathways via treatment with the amivantamab and combination TKI combination may improve overall efficacy by limiting the compensatory pathway activation.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the informed consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Participant is ≥ 18 years of age.
4. Participant has histologic or cytologic confirmation of locally advanced (unresectable) or metastatic NSCLC with a known (and documented) ALK, ROS1, or RET fusion based on approved diagnostic testing methods specified below. Not that NGS testing is required for all participants, but screening if any of the test below are positive.

   a. IHC: For ALK NSCLC only using the ALK D5F3 antibody b. FISH with ≥15% of 100 cells sampled constituting positivity c. NGS using a CLIA-certified test
5. Participants must have clinical progression on at least one prior FDA-approved TKI. They must be on a TKI at the same dose for at least 8 weeks without radiographic progression or clinical intolerance of the TKI prior to enrolling on this study. TKIs that will be considered include (but not limited to):

   1. ALK fusions - alectinib, brigatinib, lorlatinib
   2. ROS1 fusions - entrectinib, lorlatinib
   3. RET fusions - selpercatinib, pralsetinib
6. Participants must have at least 1 measurable lesion by RECIST v1.1 criteria using computed tomography (CT) scan or magnetic resonance imaging (MRI).

   1. Measurable CNS lesions ≥10mm must be captured as overall and intracranial RECIST target lesions. CNS lesions 5-9mm may be included in the intra-cranial data set alone but must be listed as non-target lesions.
   2. Measurable, treated brain metastases (≥ 10mm) growing after whole-brain radiotherapy (WBRT) or resection are allowed as target lesions, but lesions growing after stereotactic radiosurgery (SRS) are allowed as target lesions only if radiation necrosis or pseudoprogression is ruled out.
7. Participant has an Eastern Cooperative Oncology Group (ECOG) score of 0-2
8. Participant has a life expectancy of greater than 12 weeks, per investigator discretion.
9. Participant can ingest oral medications.
10. Participant has received the final dose of any of the following treatments/procedures with the specified minimum intervals before the first dose of study drug (unless in the opinion of the Sponsor-Investigator, the medication will not interfere with the study or compromise participant safety).

    Chemotherapy 21 days Antibody-drug conjugate (ADC) 28 days Immune checkpoint inhibitors (ICI) 28 days Locally ablative radiotherapy 28 days Palliative radiotherapy 14 days Major surgery 28 days
11. Participant has adequate organ function as determined by the following laboratory values.

    Absolute neutrophil count (ANC)* ≥ 1,500/mm3 (≥ 1.5 x One times ten to the ninth/L) Platelets† ≥ 75,000/mm3 (≥ 75 x One times ten to the ninth/L) Hemoglobin† ≥ 9 g/dL Renal function: Serum creatinine ≤ 1.5 x upper limit normal (ULN) OR creatinine clearance ≥50 mL/min/1.73 m2 via Cockcroft-Gault Liver transaminases (ALT/AST) ≤ 3 x ULN
    * 5 x ULN, if liver metastases are present on screening Bilirubin ≤ 1.5 x ULN
    * 3.0 x ULN, if patient has Gilbert's disease Amylase and lipase ≤ 1.5 x ULN

      * Participants cannot be receiving growth factor support using granulocyte-stimulating colony factor (G-CSF) during the screening visit.

        * Participants cannot receive transfusion support up to one week prior to the screening period.
12. Female participant of childbearing potential (defined as a sexually mature woman who has not undergone a hysterectomy [surgical removal of the uterus] or bilateral oophorectomy, or if ≥ 45 years old, has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must:

    1. Have 1 negative pregnancy test as verified by an Investigator prior to starting study therapy. This applies even if the subject practices true abstinence from heterosexual contact.
    2. Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis) or agree to use and be able to comply with a barrier method plus a hormonal method of contraception without interruption 28 days prior to starting investigational product, during the study therapy (including dose interruptions), and for 3 months after discontinuation (or longer if required by local requirements) of study therapy. The method of contraception must be a barrier method plus a hormonal method to prevent pregnancy.
    3. Participants must agree to continue contraception throughout the study and continuing through 3 months after the last dose of study drug. Note: If the childbearing potential changes after start of the study (e.g., woman who is not heterosexually active becomes active, premenarchal woman experiences menarche) the woman must begin a highly effective method of birth control, as described above.
    4. A woman of childbearing potential must have a negative serum or urine (b- human chorionic gonadotropin [b-hCG]) at Screening.
    5. A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 6 months after receiving the last dose of study drug.
    6. A female participant must agree not to be pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 3 months after the last dose of study treatment.
13. A man who is sexually active with a woman of childbearing potential must agree to use a condom with spermicidal foam/gel/film/cream/suppository and his partner must also be practicing a highly effective method of contraception (i.e., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device [IUD] or intrauterine system [IUS]). If the subject is vasectomized, he must still use a condom (with or without spermicide), but his female partner is not required to use contraception. The subject must also not donate sperm during the study and for 6 months after receiving the last dose of study drug, even if he has undergone a successful vasectomy.

Exclusion Criteria:

1. Participant has received an investigational drug within a 28-day period (or within 5 half-lives, whichever is shorter) before the first dose of study drug or is currently participating in another interventional clinical trial, unless in the opinion of the Sponsor-Investigator, the medication will not interfere with the study procedures or compromise subject safety.
2. The participant cannot have ever received an EGFR TKI (e.g. osimertinib), EGFR- directed monoclonal antibody (e.g. cetuximab), MET TKI (e.g. capmatinib, tepotinib), MET-directed monoclonal antibody (e.g. amivantamab) or MET-directed antibody-drug conjugate (e.g. telisotuzumab vedotin) prior to study entry. For patients with ALK or ROS1 NSCLC, crizotinib cannot be used within 3 months of screening.
3. Participants who have progressed on a TKI in less than 8 weeks
4. The participant has evidence of neuroendocrine differentiation or small cell transformation on the screening biopsy.
5. The patient has no evidence of an ALK, ROS1, and RET gene fusion as determined by molecular testing. Acquired resistance mechanisms detected through NGS (or FISH) testing for which alternative therapies exist may potentially be eligible after consultation with the PI.
6. Participants with active, symptomatic, central nervous system disease defined as follows:

   1. Leptomeningeal disease.
   2. Symptomatic cord compression from metastatic disease.
   3. Untreated, symptomatic brain metastases
   4. Patients with brain metastases may be potentially eligible provided that all the following criteria are met:

   i. They are not on prednisolone 20mg equivalents daily prior to enrolling in the study.

   ii. Anticonvulsants will be permitted provided the patient has been on a stable dose for a period of 2 weeks prior to Study Day 1.

   iii. Procedural interventions (such as ventriculoperitoneal shunt) greater than 12 weeks prior to Study Day 1.

   iv. Palliative radiotherapy (either whole brain radiotherapy or stereotactic radiosurgery) ≥ 28 days prior to screening.
7. Participant has active cardiovascular disease defined as the following:

   1. Congestive heart failure (CHF), defined as New York Heart Association (NYHA) class III-IV or hospitalization for CHF within 6 months of study Day 1.
   2. Symptomatic acute coronary syndrome, unstable angina, or active ischemia requiring coronary artery stenting, angioplasty, or bypass grafting within 12 weeks prior to starting investigational drug.
   3. Participant has evidence of current, uncontrolled, clinically significant, unstable arrhythmias. Participants receiving active anti-arrhythmic therapy are not eligible with the following exceptions:

   i. Participants with atrial fibrillation medically controlled for greater than 4 weeks prior to Study Day 1.

   ii. Participants who have medical pacemakers for control of arrhythmias. d. Participant has medically uncontrolled hypertension (defined as ≥ 160 mmHg systolic blood pressure (SBP) and ≥ 100 mmHg diastolic blood pressure (DBP).

   e. Clinically significant, acute deep vein thrombosis or pulmonary embolism within 6 months prior to first dose of study drug. Clinically non-significant thrombosis, such as non-obstructive catheter-associated clots or incidentally detected, asymptomatic, subsegmental pulmonary emboli are not considered exclusionary.

   f. History of cerebrovascular accident or transient ischemic attack within12 weeks of enrollment.

   g. QT interval corrected by Fridericia's Formula (QTcF) prolongation to > 470ms based on a 12-lead electrocardiogram.
8. Participant has any history of interstitial lung disease (ILD), including drug induced ILD or radiation pneumonitis requiring treatment with prolonged steroids or other immune suppressive agents that is unresolved or resolved within the last 3 months
9. Participant has clinical evidence or history of ongoing significant bowel obstruction limiting oral intake, active uncontrolled malabsorption syndromes, or any other gastrointestinal disorder or defect that would interfere with absorption, distribution, metabolism, or excretion of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity.
10. Participant has an additional primary malignancy within 2 years prior to enrollment with following exceptions:

    1. Adequately resected non-melanoma skin cancer.
    2. Superficial bladder tumors (Ta, Tis, or T1).
    3. Adequately treated intraepithelial carcinoma of the cervix uteri.
    4. Low-risk, non-metastatic prostate cancer following local treatment or ongoing active surveillance.
    5. Any other curatively treated in situ disease.
11. Participant is positive for human immunodeficiency virus (HIV), with 1 or more of the following:

    f. Receiving ART that may interfere with study treatment (consult sponsor investigator for review of medication prior to enrollment) g. CD4 count ≤ 350 at screening h. AIDS-defining opportunistic infection within 6 months of the start of screening i. Not agreeing to start ART and be on ART > 4 weeks plus having HIV viral load < 400 copies/mL at the end of 4-week period (to ensure ART is tolerated and HIV controlled).
12. Participant has active/chronic, known, untreated, hepatitis B as demonstrated by a positive hepatitis B surface antigen (HBsAg). Note: Subjects with a prior history of HBV demonstrated by positive hepatitis B core antibody are eligible if they have the following at Screening:

    j. Negative HBsAg. k. HBV DNA (viral load) below the lower limit of quantification, per local testing.

    l. Subjects with a positive HBsAg due to recent vaccination are eligible if HBV DNA (viral load) is below the lower limit of quantification, per local testing.
13. Participant has active/chronic, known, untreated, hepatitis C infection as demonstrated by a positive HCV antibody with detectable HCV viral load.

    Note: Subjects with a prior history of HCV, who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible.
14. Participant has a concurrent and uncontrolled medical illness which would preclude study conduct and assessment, including, but not limited to the following medical conditions: an active infection requiring systemic therapy, bleeding disorder, clinically unstable ophthalmologic condition, diabetes mellitus with end-organ damage, pulmonary diseases, or alcoholic liver disease.
15. Participant is a pregnant or lactating woman.
16. Participant has a history of severe allergic reactions to any of the study intervention components.
17. Participant has a medical or psychiatric condition, which might compromise their ability to give written informed consent or to comply with the study protocol visits and procedures.
18. Participant has immune-mediated rash from checkpoint inhibitors that has not resolved prior to enrollment.
19. Use of live or live-attenuated vaccines within 30 days of screening.
20. Participant has significant reversible toxicities from prior anti-cancer therapy that have not recovered to Grade 1 or baseline (higher grades of alopecia and neuropathy up to Grade 2 will be permitted).
21. Participant had major surgery excluding placement of vascular access or tumor biopsy, or had significant traumatic injury within 4 weeks before enrollment, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study. Note: Participants with planned surgical procedures to be conducted under local anesthesia may participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Determine the MTD in adult participants with advanced NSCLC | 18 months
  The MTD is defined as the dose combination with a DLT rate closest to the target DLT rate of 22%. An unevaluable patient is one who fails to complete dosing in C1 unless due to drug-related toxicities. The starting dose level will be dose level 0.
Determine the recommended phase 2 dose in adult participants with advanced NSCLC | 20 months
Estimate the objective response rate (ORR) of amivantamab in combination with common TKIs used in ALK, ROS1, and RET advanced NSCLC progressing on TKIs | 40 months
  To estimate the objective response rate (ORR) of amivantamab in combination with common TKIs used in ALK, ROS1, and RET advanced NSCLC progressing on TKIs. This will be done per investigator and independent central review via RECIST 1.1. and RANO guidelines (for patients with brain metastases)

SECONDARY OUTCOMES:
Collect treatment-related adverse events (TRAEs) | 40 months
  All graded AEs (using CTCAE 5.0 criteria)
Collect treatment-emergent adverse events | 40 months
  All graded AEs (using CTCAE 5.0 criteria)
To evaluate the overall progression free survival (PFS) in patients treated with amivantamab in combination with concurrent TKI in patients with advanced NSCLC with ALK, ROS1, and RET gene fusions | 40 months
To evaluate the intracranial progression free survival (PFS) in patients treated with amivantamab in combination with concurrent TKI in patients with advanced NSCLC with ALK, ROS1, and RET gene fusions | 40 months
To evaluate the extracranial progression free survival (PFS) in patients treated with amivantamab in combination with concurrent TKI in patients with advanced NSCLC with ALK, ROS1, and RET gene fusions | 40 months
To evaluate the overall disease control rate (DCR) among patients treated with amivantamab in combination with concurrent TKI in patients with advanced NSCLC with ALK, ROS1, and RET gene fusions. | 40 months
To evaluate the intracranial disease control rate (DCR) among patients treated with amivantamab in combination with concurrent TKI in patients with advanced NSCLC with ALK, ROS1, and RET gene fusions. | 40 months
To evaluate the extracranial disease control rate (DCR) among patients treated with amivantamab in combination with concurrent TKI in patients with advanced NSCLC with ALK, ROS1, and RET gene fusions. | 40 months
To evaluate the overall duration of response (DOR) among responders in patients treated with amivantamab in combination with concurrent TKI in patients with advanced NSCLC with ALK, ROS1, and RET gene fusions | 40 months
To evaluate the intracranial duration of response (DOR) among responders in patients treated with amivantamab in combination with concurrent TKI in patients with advanced NSCLC with ALK, ROS1, and RET gene fusions | 40 months
To evaluate the extracranial duration of response (DOR) among responders in patients treated with amivantamab in combination with concurrent TKI in patients with advanced NSCLC with ALK, ROS1, and RET gene fusions | 40 months

CONTACTS AND LOCATIONS:
Overall Officials: Erin Schenk, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - City of Hope Cancer Center, Duarte, California
  - Outpatient CTRC, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No